CLINICAL TRIAL: NCT01860794
Title: Investigator Clinical Trial for Evaluation of Safety and Tolerability After Transplantation of Fetal Mesencephalic Dopamine Neuronal Precursor Cells in Patients With Parkinson's Disease
Brief Title: Evaluation of Safety and Tolerability of Fetal Mesencephalic Dopamine Neuronal Precursor Cells for Parkinson's Disease
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bundang CHA Hospital (Other)
Responsible Party: Principal Investigator, Sang Sup Chung, Professor, Bundang CHA Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PBC09-074
Record Dates: First submitted 2013-05-14; First posted 2013-05-23 (Estimated); Last update posted 2020-07-10 (Actual); Status verified 2020-07

CONDITIONS: Idiopathic Parkinson Disease; Primary Parkinsonism
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Mesencephalic Neuronal Precursor Cells (Other)
  Interventions: Drug: Mesencephalic Neuronal Precursor Cells

INTERVENTIONS:
Drug: Mesencephalic Neuronal Precursor Cells — All the patients are continuously registered for this study. Data monitoring committee inspects the clinical results of first patient and decides whether the treatment for four subjects are appropriate to proceed. 5 subjects of each group are subject to inspection by Data monitoring committee after the end of tracking fifth patients.

SUMMARY:
The purpose of clinical trials is to evaluate safety and tolerability of Fetal Mesencephalic Dopamine Neuronal Precursor Cells as a treatment for Patients with Parkinson's disease.

DETAILED DESCRIPTION:
This study is phase I/II clinical trials which is accessible to those involved in the study and conducted by only Bundang CHA hospital.

The progress of the clinical trails is reported to and evaluated by Data monitoring committee before the enrolment of next human subject.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients with idiopathic or primary Parkinson's disease
2. Hoehn and Yare (HY) stage III or IV
3. more than 33% improvement Part III UPDRS score after one injection of levodopa in the morning
4. Patients aged less than 70
5. Great decrease of dopamine uptake in putamen, particularly posterior part, in Positron emission tomograph(PET) before surgery

Exclusion Criteria:

1. Atypical or secondary parkinsonism
2. Medical history of severe depression with Beck Depression Inventory(BDI) scores greater than 30
3. Psychological disorders (illusion, delusion, schizophrenia)
4. Dementia with K-MMSE(Korean mini-mental state examination) scores less than 24
5. Epilepsy
6. Medial history of brain surgery
7. Medical history of other brain diseases
8. Hemorrhagic tendency
9. Severe internal diseases such as poor general condition, hypertension, chronic respiratory disease, ischemic heart disease, cancer
10. Experience of participating in clinical trial within 30 days
11. Female patients who have the chances of getting pregnant during clinical trial and do not use the approved birth controls
12. Pregnant or lactating women
13. Patients who are not considered to be eligible to participate in clinical trial

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2013-05; Primary Completion 2022-04 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Presence or absence of cancer foramtion and infection | 5 years
  If not included in the following criteria, the cells are are considered to be safe and tolerable.
  * Cells with grade 3 or more in NCI grading system
  * Cells contaminated with infectious materials
  * Cells with risk of cancer formation

SECONDARY OUTCOMES:
Score of Unified Parkinson's Disease Rating Scale (UPDRS) | 5 years
  UPDRS, most commonly used, is designed to assess the severity of parkinson's disease, making the quantitative measurement of the extent. Part III of UPDRS corresponds to motor evaluation and is the most reliable for detecting symptomatic progression.
  UPDRS improvement ratio(%) = ((the value of UPDRS before surgery - the value of UPDRS after surgery) / (the value of UPDRS before surgery)) X 100
Detection of positron emission in Putamen using Positron emission tomograph(PET) | 5 years
  In pet analysis, putamen activity is investigated via radioactivity before cell transplantation and 12,24,36,48,60 months after the treatment.
Dyskinesia scale scores(CAPSIT-PD) | 5 years
  Overall inspection was carried out before transplantation and 1, 3, 6, 9, 12, 15, 18, 21, 24, 30, 36, 42, 48, 54, 60 months after the treatment for determining whether the cells have therapeutic effects.
Pronation-supination test, Hand/Arm movement between two points, finger dexterity, stand-walk-sit-test | 5 years
  Comprehensive clinical assessment for examining the improvements in self reporting and timed testing before the cell transplantation and 1, 3, 6, 9, 12, 15, 18, 21, 24,30, 36, 42, 48, 54, 60 months after the treatment:Pronation-supination test, Hand/Arm movement between two points, finger dexterity, stand-walk-sit-test.
Score of activity of daily living (ADL) scale | 5 years
  Comprehensive clinical assessment for examining the improvements in activity of daily living before the cell transplantation and 1, 3, 6, 9, 12, 15, 18, 21, 24,30, 36, 42, 48, 54, 60 months after the treatment.
Score of Korean mini-mental examination (K-MMSE) | 5 years
  Comprehensive clinical assessment for examining the improvements in mental state before the cell transplantation and 1, 3, 6, 9, 12, 15, 18, 21, 24,30, 36, 42, 48, 54, 60 months after the treatment.
Motor fluctuation scale scores | 5 years
  Comprehensive clinical assessment for identifying the presence of motor fluctuation symptoms before the cell transplantation and 1, 3, 6, 9, 12, 15, 18, 21, 24,30, 36, 42, 48, 54, 60 months after the treatment.
Satisfaction score with patient questionnaire | 5 years
  Measure of patient satisfaction before the cell transplantation and 1, 3, 6, 9, 12, 15, 18, 21, 24,30, 36, 42, 48, 54, 60 months after the treatment.
Dopaminergic drug dose | 5 years
  Measure of dopaminergic drug dose before the cell transplantation and 1, 3, 6, 9, 12, 15, 18, 21, 24,30, 36, 42, 48, 54, 60 months after the treatment.
Tremor, postural instability, motor dysfunction, gait disturbance | 5 years
  Using video recording, assessment for symptoms such as tremor, postural instability, motor dysfunction and gait disturbance before the cell transplantation and 1, 3, 6, 9, 12, 15, 18, 21, 24,30, 36, 42, 48, 54, 60 months after the treatment.
Assessing the extent of recovery with patient's diary | 5 years
  Assessing the extent of recovery based on patient's diary before the cell transplantation and 1, 3, 6, 9, 12, 15, 18, 21, 24,30, 36, 42, 48, 54, 60 months after the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Sang Sup Chung, M.D., Ph.D., Principal Investigator — CHA University
Locations (1):
- CHA Bundang Medical Center, CHA University, Seongnam-si, Gyeonggi-do, South Korea